CLINICAL TRIAL: NCT03892876
Title: Pilot Trial of Stimulus-response Potentiation in Schizophrenia
Brief Title: Trial of Stimulus-response Potentiation in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kyrillos Meshreky, Assistant lecturer of Psychiatry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-173-2019
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Schizophrenia TS+ve (Experimental): Schizophrenia patients who receive auditory high frequency Tetanizing Stimulation
  Interventions: Diagnostic Test: Auditory High Frequency Tetanizing Stimulation
- Schizophrenia TS-ve (Sham Comparator): Schizophrenia patients who receive sham comparator
  Interventions: Diagnostic Test: Sham Comparator
- Control TS+ve (Experimental): Healthy controls who receive auditory high frequency Tetanizing Stimulation
  Interventions: Diagnostic Test: Auditory High Frequency Tetanizing Stimulation
- Control TS-ve (Sham Comparator): Healthy controls who receive sham comparator
  Interventions: Diagnostic Test: Sham Comparator

INTERVENTIONS:
Diagnostic Test: Auditory High Frequency Tetanizing Stimulation — 50 ms tone pips presented at high frequency for 120 seconds
  Arms: Control TS+ve; Schizophrenia TS+ve
Diagnostic Test: Sham Comparator — auditory tone pips with interstimulus interval (ISI) 1 sec
  Arms: Control TS-ve; Schizophrenia TS-ve

SUMMARY:
This clinical trial aims at examining the effects of auditory high-frequency stimulation in schizophrenia patient, aiming to increase their AEPs, which are known to be attenuated from previous literature

DETAILED DESCRIPTION:
Schizophrenia is a chronic psychiatric disorder with a lifetime prevalence of 4.0 per 1,000. The introduction of antipsychotic medications in the 1950s resulted in marked clinical improvement in the symptom profile of schizophrenia, nevertheless the disease still contributes to a significant proportion of global disease burden in terms of both morbidity and mortality. In this regard, cognitive deficits and residual negative symptoms are considered major contributing factors to psychosocial disability and poor functional outcome associated with the disorder.

Higher-order cognitive functions; e.g. working memory and executive functions; show variable deficits and are considered a core clinical symptom of schizophrenia. On the other hand, the disorder is also characterized by abnormalities at the basic level of primary sensory processing, i.e. auditory, visual and somatosensory processing. Such abnormalities in the primary process of sensory perception could change the sensory experiences of schizophrenia patients and thus contribute to the psychopathology.

Event-related potentials (ERPs) are the neurophysiological correlates of sensory processing. ERP abnormalities have been widely described in schizophrenia literature: Pre-pulse inhibition of startle (PPI) in which a weaker pre-stimulus (pre-pulse) inhibits the reaction to a subsequent strong startling stimulus (pulse) is impaired in schizophrenia. P50 suppression, a measure of sensory gating, is also often absent or reduced in the disorder. N100; a measure of basic auditory sensory perception; shows significant amplitude reduction in patients compared to controls. Mismatch negativity (MMN), a measure of automatic deviance detection and shows characteristic attenuation in schizophrenia. P300, which is involved in higher-level stimulus evaluation and categorization, also shows abnormalities along the disease course.

In the study by Clapp et al., 2005, auditory high frequency stimulation (tetanizing stimulation) resulted in an increase in auditory-evoked potentials (AEPs) in healthy individuals; i.e. an increase in N1 amplitude that persisted even after stimulation. This augmentation of N1 amplitude was regarded as a result of plastic synaptic potentiation similar to long-term potentiation (LTP) described after electrical tetanic stimulation in cellular studies. Similar findings were later replicated by Lei et al., 2017, where they used pure tones, narrow band noises and white noise to induce stable potentiation and augmentation of N1 amplitude.

ELIGIBILITY:
For Schizophrenia group:

Inclusion Criteria:

* Able to give written informed consent
* Males (ages 20-50 years)
* Diagnosis of schizophrenia as confirmed by Structured Clinical Interview for DSM-V-TR (SCID)
* on stable doses of antipsychotic medications for at least 15 days
* scores 4 or more on at least one item of the Positive and Negative Syndrome Scale.

Exclusion Criteria:

* History of / or current medical/neurological illnesses e.g. mental retardation (DSM-V) or epilepsy or significant head trauma
* Any type of hearing deficit will be excluded by audiometry assessment
* Substance abuse in the past 2 months
* medical conditions that make it difficult for the patient to visit the clinic in the designed schedule.

For control group:

Inclusion criteria:

* able to give written informed consent
* males (ages 20-50).

Exclusion criteria:

* History of / or current medical/neurological illnesses e.g. mental retardation (DSM-V) or epilepsy or significant head trauma
* Any type of hearing deficit
* if they meet any axis-I diagnosis according to DSM-V confirmed by SCID.
* scores 2 or more on one item of the Positive and Negative Syndrome Scale

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
N100 wave (AEP) amplitude in µv [microvolts] | 1-2 hours
  N100 or N1 is a large, negative-going evoked potential measured by electroencephalography. It peaks in adults between 80 and 120 milliseconds after the onset of a stimulus, and distributed mostly over the fronto-central region of the scalp.
P300 wave amplitude in µv [microvolts] (auditory odd-ball task) | 1-2 hours
  The P300 (P3) wave is an event related potential (ERP) component elicited in the process of decision making. It is considered to be an endogenous potential, as its occurrence links not to the physical attributes of a stimulus, but to a person's reaction to it. More specifically, the P300 is thought to reflect processes involved in stimulus evaluation or categorization.

SECONDARY OUTCOMES:
performance of Wisconsin Card Sorting test (WCST). | 3 days
  Wisconsin Card Sorting Test (WCST) is a neuropsychological test of "set-shifting", i.e. the ability to display flexibility in the face of changing schedules of reinforcement.

CONTACTS AND LOCATIONS:
Overall Officials: Ola O Shahin, MD, Study Director — Department of Psychiatry-University of Cairo; Vishwajit L Nimgaonkar, PhD, Study Director — Department of Psychiatry-University of Pittsburgh
Locations (1):
- Department of Psychiatry-Faculty of medicine-University of Cairo, Cairo, Cairo Governerate, Egypt